CLINICAL TRIAL: NCT00002266
Title: An Open Parallel Study to Determine the Optimum Dosing Schedule for AS-101 in AIDS/ARC Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 045B; 753A-103-US
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1990-12

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; ammonium trichloro(dioxoethylene-O,O'-)tellurute
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — ammonium trichloro(dioxoethylene-O,O'-)tellurate

INTERVENTIONS:
Drug: AS-101

SUMMARY:
To compare AS-101 dosing schedules (once a week; 3 times a week; 5 times a week; or 5 times per week on alternate weeks) on the effect on clinical immunology and virus burden in AIDS or AIDS related complex (ARC) patients.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Standard therapy for infections.
* Acyclovir.
* Ganciclovir.
* Allowed only with permission of Wyeth-Ayerst medical monitor:
* Zidovudine (AZT).
* Immunomodulators.
* Specific therapy for malignancies (including Kaposi's sarcoma).

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Evidence of severe liver dysfunction (serum albumin < 3 g/dl, SGOT or SGPT > 5 x upper limit of normal, prothrombin time > 15 seconds), or gastrointestinal, renal, respiratory, endocrine, hematologic, cardiovascular system abnormalities or psychiatric disorder other than abnormalities secondary to AIDS or AIDS related complex (ARC).
* Evidence of AIDS-related central nervous system involvement.
* Disseminated Kaposi's sarcoma.

Concurrent Medication:

Excluded without permission of Wyeth-Ayerst medical monitor:

* Zidovudine (AZT).
* Immunomodulators.
* Specific therapy for malignancies (including Kaposi's sarcoma).

Patients with the following are excluded:

* Evidence of major system abnormalities other than abnormalities secondary to AIDS or AIDS related complex.
* Concomitant conditions as specified in Patient Exclusion Co-existing Conditions.
* Unlikely or unable to comply with the requirements of the protocol.

Prior Medication:

Excluded within 4 weeks of study entry:

* Systemic antiviral agents.
* Immunosuppressive agents.
* Immune stimulators such as BCG vaccine, isoprinosine, or other immunomodulators.

Patients must:

* Have a diagnosis of AIDS or AIDS related complex (ARC).
* Demonstrate intolerance or refusal to take zidovudine (AZT).
* Provide written informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Univ of Arizona / Health Science Ctr, Tucson, Arizona, United States